CLINICAL TRIAL: NCT02637895
Title: Evaluation of the Efficacy of Vortioxetine for Posttraumatic Stress Disorder
Brief Title: Vortioxetine for Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Takeda (Industry); Emory University (Other)
Responsible Party: Principal Investigator, Philip D. Harvey, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20150534
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD,; trauma; stress disorder; post-traumatic stress disorder; anxiety disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Stress Disorders, Traumatic; Anxiety Disorders | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo pill once daily for 12 weeks of active treatment.
  Interventions: Drug: Placebo
- Vortioxetine (Active Comparator): Vortioxetine pill 10mg once daily up to 4 weeks followed by 20mg once daily if tolerated for the rest of the study. Patients unable to tolerate the 20 mg/day dose may be reduced to 10 mg/day between weeks 4 and 8. The dose of study medication should remain stable for weeks 8-12.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Placebo — Placebo pill matching Vortioxetine.
  Arms: Placebo
Drug: Vortioxetine — Immediate Release 10 mg. Vortioxetine Pill
  Arms: Vortioxetine

SUMMARY:
Post-traumatic stress disorder (PTSD) can result from having experienced or witnessed a traumatic event. Patients with PTSD symptoms can sometimes experience symptom relief after treatment with antidepressants; however, few patients experience complete symptom relief. There is a need to develop new treatments for PTSD.

This study will evaluate if 12 weeks of using Vortioxetine relieves PTSD symptoms. Vortioxetine has been approved for the treatment of depression; however, Vortioxetine has not been approved by the Food and Drug Administration for the treatment of PTSD.

DETAILED DESCRIPTION:
Patients included in the study will either take the study medication or will take a placebo, a pill without the active medication. This will be determined by chance like a flip of a coin.

Study procedures will include taking study medication and coming to regular in-clinic visits. Depending on the study visit, study tests may include the following: medical evaluations, physical exams, body measurements, vital signs, blood and urine tests, pregnancy tests, genetic testing, heart function monitoring, clinical and psychiatric measures, neuropsychological testing (for example, investigators will test how well you remember words or how fast you perform a certain task), a function test (for example, investigators will test how well you perform certain daily tasks), and a test to measure your startle response. A startle response is an unexpected response by a sudden activity.

ELIGIBILITY:
Inclusion

1. Males and Females between the ages of 18 and 65
2. Fulfills Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for primary diagnosis of PTSD.
3. Able to give consent
4. Willingness to sign the treatment contract
5. A negative urine toxicology
6. For females of reproductive age, use of an effective birth control method* for the duration of the study or abstinence.
7. Duration of illness of PTSD for at least 3 months
8. An initial score at Screening, and Visit 3 (randomization) of ≥ 50 on the Clinician Administered PTSD Scale (CAPS) for PTSD Studies

Exclusion

1. Lifetime or current diagnosis of schizophrenia or other psychotic disorder, dementia, bipolar disorder.
2. Subject is currently participating in another clinical trial in which s/he is or will be exposed to an investigational or non-investigational drug or device, or has done so within the preceding month.
3. Current evidence or history of significant unstable medical illness or organic brain impairment, including stroke, Central Nervous System (CNS) tumor, demyelinating disease, cardiac, pulmonary, gastrointestinal, renal or hepatic impairment that would likely interfere with the action, absorption, distribution, metabolism, or excretion of Vortioxetine. History of moderate or more severe Traumatic Brain Injury (TBI) will also be exclusionary.
4. Patients who in the investigator's judgment pose a current suicidal or homicidal risk
5. DSM-5 substance abuse or dependence within the past 90 days. Subject has a positive urine toxicology test for illegal substances.
6. Diagnosis of anorexia nervosa, bulimia, or Obsessive Compulsive Disorder (OCD) in the past year.
7. Subject has a documented history of hepato-biliary disease including a history of, or positive laboratory results for hepatitis (hepatitis B surface antigen and/or hepatitis C antibody), and clinically significant hepatic enzyme elevation, including any one of the following enzymes greater than 3 times the upper limit of normal (ULN) value (Alanine transaminase (ALT), aspartate aminotransferase (AST), alkaline phosphatase( ALP)), or total or direct bilirubin > 1.5 x ULN, unless consistent with presumed or diagnosed Gilbert's disease
8. Subject has taken systemic corticosteroids within 2 weeks of the Randomization Visit
9. Treatment with any other psychoactive medication within 2 weeks of Visit 1, including all antidepressants, psychoactive herbal or nutritional treatment (St Johns Wort,S-Adenosyl methionine(SAM-e)), lithium, other mood stabilizers, oral antipsychotics, depot antipsychotics within 12 weeks, beta blockers, thioridazine, pimozide, opiates, anxiolytics, and sedatives (with the exception of zolpidem, eszopiclone, and zaleplon). Also any treatment with any medication that the PI judges not acceptable for this study.
10. Pregnancy or lactation*
11. Subjects who, in the opinion of the investigator, would be noncompliant with the visit schedule or study procedures (e.g. illiteracy, planned vacations, or planned hospitalizations during the study).
12. Any laboratory abnormality that in the investigator's judgment is considered to be clinically significant
13. Patients who are receiving exposure-based psychotherapy that targets PTSD symptoms
14. Current or planned litigation or other actions related to secondary gain regarding the traumatic event
15. Subject has clinical evidence of, or ElectroCardiogram (ECG) results indicating any of the following at either screen or Randomization Visit unless repeat ECG shows that the parameter had returned to within normal range by the Randomization Visit:

    * Q to T interval change (QTc)> 450 msec for men, or > 475 msec for women;
    * any cardiac condition or ECG evidence that the investigator feels may pose a potential safety concern.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Harvey, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guidetti C, Feeney A, Hock RS, Iovieno N, Hernandez Ortiz JM, Fava M, Papakostas GI. Antidepressants in the acute treatment of post-traumatic stress disorder in adults: a systematic review and meta-analysis. Int Clin Psychopharmacol. 2025 May 1;40(3):138-147. doi: 10.1097/YIC.0000000000000554. Epub 2024 Jun 14. PMID 38869978
- [Derived] Dunlop BW, Rakofsky JJ, Newport DJ, Mletzko-Crowe T, Barone K, Nemeroff CB, Harvey PD. Efficacy of Vortioxetine Monotherapy for Posttraumatic Stress Disorder: A Randomized, Placebo-Controlled Trial. J Clin Psychopharmacol. 2021 Mar-Apr 01;41(2):172-179. doi: 10.1097/JCP.0000000000001363. PMID 33587394

RESULTS

PARTICIPANT FLOW:
Groups:
- Vortioxetine: Vortioxetine pill 10mg once daily up to 4 weeks followed by 20mg once daily if tolerated for the rest of the study. Patients unable to tolerate the 20 mg/day dose may be reduced to 10 mg/day between weeks 4 and 8. The dose of study medication should remain stable for weeks 8-12.
  Vortioxetine: Vortioxetine pill 10mg once daily up to 4 weeks followed by 20mg once daily if tolerated for the rest of the study. Patients unable to tolerate the 20 mg/day dose may be reduced to 10 mg/day between weeks 4 and 8. The dose of study medication should remain stable for weeks 8-12.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine
Started | 21 | 20
Completed | 15 | 17
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 4 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Abnormal baseline lab | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.0) | 44.3 (11.9) | 42.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change Clinician Administered PTSD Scale Score
Description: Clinician-Administered PTSD Scale (CAPS-5) has a total score ranging from 0-80 with the higher score indicating greater degree of PTSD symptom severity.
Time Frame: Baseline, Up to Week 12
Population: Mixed Model Repeated Measures (MMRM) Analysis of all Intent To Treat (ITT) cases
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 21 | 20
score on a scale | 16 (3.00) | 17 (2.70)

2. Secondary Outcome: Number of Participants That Achieve Treatment Response Via Clinician Administered PTSD Scale (CAPS)-5
Description: Number of participants that achieve treatment response will be reported as those that has achieved a 30% improvement in their CAPS-5 total score from baseline. CAPS-5 has a total score ranging from 0-80 with the higher score indicating greater degree of PTSD symptom severity. Observed cases only.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 15 | 17
Participants | 9 | 11

3. Secondary Outcome: Change in Depressive Symptoms in PTSD
Description: Montgomery-Asberg Depression Rating Scale (MADRS) has a total score ranging from 0-60, with 0 meaning no depressive symptoms and 60 meaning severe depressive symptoms.(MADRS). From the total score 0-60, with 0 meaning no depressive symptoms and 60 meaning severe depressive symptoms.
Time Frame: Baseline, Up to Week 12
Population: Mixed Model Repeated Measures (MMRM) Analysis of all Intent To Treat (ITT) cases
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 21 | 20
score on a scale | 9.73 (1.95) | 12.06 (2.27)

4. Secondary Outcome: Number of Participants That Achieve Treatment Response Via CGI-I
Description: Clinical Global Impression of Improvement (CGI-I) is a 7 point Likert-scale questionnaire assessing PTSD symptoms improvement. A score of 1 indicates very much improved, 4 indicates no change and 7 indicates much worse. Treatment response will be reported as the number of participants with an improvement of 1-2 points on their CGI-I score from baseline. Analysis includes observed cases only.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 15 | 17
Participants | 10 | 11

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Only treatment-related adverse events, as evaluated by treating physician, will be reported at the 5% reporting threshold.
Arm/Group | Placebo | Vortioxetine
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 11/21 | 15/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Vortioxetine (N=20)
Diarrhea (Gastrointestinal disorders) | 4 (10) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (3) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (6) | 10 (16)
Headache (General disorders) | 4 (11) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT02637895/Prot_SAP_000.pdf